CLINICAL TRIAL: NCT03438214
Title: Effect of Intermittent Infusion Versus Continuous Infusion of Vancomycin on Kidney Failure in Critically Ill Patients: Randomized and Controlled Multicenter Clinical Trial.
Brief Title: Effect of Intermittent Infusion Versus Continuous Infusion of Vancomycin on Kidney Failure in Critically Ill Patients
Acronym: ETERNITY
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Juliano P Almeida, MD, PhD, Research associate, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 81226617.8.1001.0065
Record Dates: First submitted 2018-02-05; First posted 2018-02-19 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Gram-Positive Bacterial Infections; Nephrotoxicity; Sepsis
Keywords: Vancomycin infusion; critical ill patients; MRSA
MeSH Terms: conditions — Gram-Positive Bacterial Infections; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vancomycin continuous infusion (Active Comparator): Continuous infusion of vancomycin
  Interventions: Drug: Vancomycin Continuous infusion
- Vancomycin intermittent infusion (Active Comparator): Intermittent infusion of vancomycin
  Interventions: Drug: Vancomycin Intermittent infusion

INTERVENTIONS:
Drug: Vancomycin Continuous infusion — Will be administered a loading dose of 25mg/kg followed of 2g infused in 24h. Serum levels will be measured after the end of the loading dose (peak) and after 24 hours (steady state). The doses will be adjusted according to serum levels (between 15 and 20 mg / L) and area under curve (AUC) /MIC≥400mg.h/L
  Other Names: Continuous infusion
  Arms: Vancomycin continuous infusion
Drug: Vancomycin Intermittent infusion — Will be administered a loading dose of 25mg/kg followed of 1g every 12h. Serum levels will be measured after the end of the loading dose (peak) and one hour before the next dose (trough). The doses will be adjusted according to serum levels (between 15 and 20 mg / L) and AUC/MIC≥400mg.h/L.
  Other Names: Intermittent infusion
  Arms: Vancomycin intermittent infusion

SUMMARY:
This is a randomized, controlled multicenter clinical trial. The purpose of this study is to compare the continuous infusion of vancomycin with intermittent infusion regarding the effectiveness to reach the target serum level and the relationship between infusion type and nephrotoxicity in critically ill patients.

DETAILED DESCRIPTION:
The vancomycin is a glycopeptide antimicrobial which has been used for 50 years against gram-positive microorganisms and remains effective against multiresistant bacteria as the methicillin resistant Staphylococcus aureus (MRSA), the main microorganism causing nosocomial infections. Around the world, the continuous infusion of vancomycin has been studied and associated with less rate of nephrotoxicity. This is a randomized, controlled multicenter clinical trial that will compare continuous infusion with the intermittent vancomycin infusion, the relationship between infusion type with rate of nephrotoxicity and the time to target therapeutic serum in critically ill patients at the intensive care units of the Cancer Institute of the State of Sao Paulo (ICESP) and the Heart Institute (Incor).

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients
* Treatment with vancomycin
* Preserved renal function.

Exclusion Criteria:

* Cystic fibrosis
* Chronic renal failure
* Acute renal failure
* Having received vancomycin in the last 24 hours
* Vancomycin hypersensibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2018-04-28 (Estimated); Primary Completion 2020-02-28 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Acute renal failure | 30 days after randomization
  Acute renal failure stage 1 according criteria AKIN (Acute Kidney Injury Network).

SECONDARY OUTCOMES:
Acute renal failure | 30 days after randomization
  Acute renal failure stages 2 or 3 according criteria AKIN (Acute Kidney Injury Network).
Hypersensibility reactions with vancomycin | 30 days after randomization
  Skin rash, bronchospasm or anaphylaxis / anaphylactic shock.
Length of ICU stay | 30 days after randomization
  Therapeutic efficacy with less length of ICU stay
Time of treatment with the antimicrobial | 30 days after randomization
  Therapeutic efficacy with less time of treatment with the antimicrobial
Length of hospitalization | 30 days after randomization
  Therapeutic efficacy with less length of hospitalization
Mortality rate | 30 days after randomization
  Therapeutic efficacy with less mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Juliano P Almeida, Professor, Principal Investigator — University os São Paulo; Estela M de Oliveira, PhD student, Principal Investigator — University os São Paulo
Locations (1):
- Faculty of Medicine University os São Paulo, São Paulo, São Paulo, Brazil